CLINICAL TRIAL: NCT05872841
Title: Efficacy and Safety of Recombinant Human Adenovirus Type 5 Injection in Combination With TACE-based Combination Therapy in Patients With Stage IIIa Primary Hepatocellular Carcinoma With Portal Vein Thrombosis
Brief Title: H101 Combined With TACE for Primary Hepatocellular Carcinoma With Portal Vein Thrombosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2023-0009
Record Dates: First submitted 2023-04-23; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-07

CONDITIONS: Primary Hepatocellular Carcinoma; Portal Vein Thrombosis
Keywords: recombinant human adenovirus type 5; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human adenovirus type 5 combined with TACE (Experimental): Recombinant human adenovirus type 5: The recombinant human adenovirus type 5 injection is administered intratumorally 48-72h prior to TACE treatment. The recombinant human adenovirus type 5 injection was diluted to 30% of the total tumor volume with saline before administration.
  TACE: Chemotherapeutic drugs were specifically oxaliplatin 85 mg/m2, calcium folinic acid 400 mg/m2, 5-fluorouracil 1200 mg/m2, and then superfluid iodinated oil bolus was given according to the intraoperative imaging tumor blood supply.
  Interventions: Drug: Recombinant human adenovirus type 5 + TACE

INTERVENTIONS:
Drug: Recombinant human adenovirus type 5 + TACE — 1. Recombinant human adenovirus type 5 : Recombinant human adenovirus type 5 injection is administered intratumorally 48-72h prior to TACE treatment.Before administration, the recombinant human adenovirus type 5 injection was diluted to 30% of the total tumor volume with normal saline. H101 dose:
     ① The sum of the maximum diameters of the lesions was ≤10cm, and the total dose was 1. 0×1012vp (2 injections);
     ② The sum of the maximum diameters of the lesions was >10cm, and the total dose was 1. 5×1012vp (3 injections);
  2. TACE：The specific chemotherapeutic drugs were: oxaliplatin 85mg/m2, calcium folinic acid 400mg/m2, 5-fluorouracil 1200mg/m2, followed by superfluid iodinated oil bolus according to the intraoperative contrast tumor blood supply.
  Recombinant human adenovirus type 5 was administered in combination with TACE in cycles of every 3 weeks for a total of 2-4 cycles.
  Other Names: H101+TACE

SUMMARY:
This study is the first to compare the efficacy and safety of recombinant human adenovirus type 5 injection via hepatic artery infusion combined with TACE-based combination therapy for the treatment of patients with stage IIIa primary hepatocellular carcinoma with portal vein carcinoma thrombosis, providing a safe and reliable treatment method for the clinical treatment of this group of patients, and also providing a reference and basis for the treatment of other tumors with this new treatment model.

DETAILED DESCRIPTION:
This is a prospective, single-arm study to evaluate the efficacy and safety of recombinant human adenovirus type 5 injection combined with TACE-based combination therapy in patients with stage IIIa primary hepatocellular carcinoma with portal vein carcinoma thrombosis. Subjects will be examined and evaluated at the study center, and after meeting the inclusion criteria, patients will be enrolled in a combination of recombinant human adenovirus type 5 injection via hepatic artery infusion and TACE regimen. The study is divided into screening period, baseline period, treatment period, and follow-up period. Follow-up after the end of treatment will be every 3 months until death or the end of this study. The primary study endpoint of this study is disease control rate (DCR) (up to 1 year), while progression free survival (PFS) (up to 1 year), 1-year overall survival rate, and distant metastasis rate are observed, and adverse events occurring during the study period are monitored for safety Data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years, regardless of gender;
2. Patients with stage IIIa primary liver cancer diagnosed by histology or imaging;
3. ECOG physical status score of 0-1;
4. Expected survival time ≥ 3 months;
5. Received no liver protective and supportive treatment within two weeks before enrollment, and met the following conditions:

   * White blood cell count ≥3.0×109/L, neutrophil absolute value ≥3.0×109/L, platelet count ≥50×109/L, hemoglobin > 100g/L;
   * INR≤1.5 and APTT≤1.5 upper limit of normal or partial prothrombin time (PTT) ≤1.5 upper limit of normal;
   * Total bilirubin (TBIL) ≤2.5 times the upper limit of normal value; ALT and AST≤5 times the upper limit of normal value; Serum creatinine ≤1.5 times the upper limit of normal value;
   * Creatinine clearance ≥50ml/min.
6. Voluntary participation in this study and signing of the informed consent form;
7. Female patients of childbearing age or male patients whose sexual partners are women of childbearing age are required to use effective contraception throughout the treatment period and for 6 months after the last dose.

Exclusion Criteria:

1. Pregnant or lactating women, men or women who do not wish to use effective contraception;
2. Patients who have received previous treatment with lysoviruses (e.g., T-VEC), interventional therapy, or TACE;
3. Those who are being treated with antiviral drugs;
4. having received any other experimental drug, antimicrobial drug, or participated in another interventional clinical trial within 4 weeks prior to enrollment
5. Those with a known allergy to the study drug or its active ingredient, or a history of allergy to similar biological agents
6. Evidence of Child-Pugh C hepatic function or hepatocellular dysregulation, including those with refractory ascites, ruptured esophageal or gastric variceal bleeding, and hepatic encephalopathy
7. presence of a history of immunodeficiency or autoimmune disease or long-term systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to enrollment
8. With any unstable systemic disease, including but not limited to: severe infection, hypertensive patients, uncontrolled diabetes mellitus, unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia, abnormal mental status or active cerebral hemorrhage, myocardial infarction, congestive heart failure, severe arrhythmias requiring drug therapy, renal or metabolic disease, severe hepatic dysfunction (including severe jaundice, hepatic encephalopathy, refractory ascites or hepatorenal syndrome), multiple organ failure with renal dysfunction;
9. Previous or concurrent other malignancies;
10. Combined medical contraindications that preclude any contrast-enhanced imaging (CT or MRI);
11. Other conditions that, in the judgment of the investigator, make the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
disease control rate (DCR) | Up to 1 year
  The percentage of patients whose tumors shrank or stabilized and remained for a certain period of time, including cases in complete remission (CR), partial remission (PR), and stable (SD)

SECONDARY OUTCOMES:
progress free survival(PFS) | Up to 1 year
  The time between the start of randomization and the onset of (any aspect of) tumor progression or death (from any cause)
overall survival(OS) | Up to 1 year
  The time from randomization to death (from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Tongguo Si, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05872841/Prot_000.pdf